CLINICAL TRIAL: NCT04969471
Title: An Interventional, Prospective, Randomized, Multi-Center, Assessor-Blinded Study Designed to Assess the Safety and Effectiveness of the EnVast Coronary Thrombectomy System As an Adjunctive Measure to Conventional Intervention in Subjects Presenting with ST-segment Elevation Myocardial Infarction (STEMI)
Brief Title: NATURE (EnVast As an Adjunct PPCI in Subjects Presenting with STEMI)
Acronym: NATURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vesalio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS-008
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Segment Elevation Myocardial Infarction (STEMI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thrombectomy Arm (Experimental): enVast stent deployed at occlusion site as first measure to obtain reperfusion and withdraw the clot
  Interventions: Device: enVast stent
- Conventional Treatment Arm (Experimental): Treatment strategies may include balloon angioplasty, manual aspiration thrombectomy and/or coronary stenting.
  Interventions: Procedure: conventional treatment

INTERVENTIONS:
Device: enVast stent — In addition to conventional treatment, the treating physician will deploy as the first measure to obtain reperfusion, a enVast stent at the occlusion site in order to withdraw the clot.
  Arms: Thrombectomy Arm
Procedure: conventional treatment — Treatment strategies may include balloon angioplasty, manual aspiration thrombectomy and/or coronary stenting.
  Arms: Conventional Treatment Arm

SUMMARY:
This study is designed to compare the safety and effectiveness of blood clot (thrombus) removal in subjects presenting with ST-segment elevation myocardial infarction (STEMI) with the enVast coronary system versus conventional intervention.

DETAILED DESCRIPTION:
A prospective, multi-center, randomized clinical trial designed to assess the safety and effectiveness of the enVast coronary thrombectomy system as an adjunctive measure to conventional intervention in subjects presenting with ST-segment elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Chest pain for > 20 min with an electrocardiographic ST-segment elevation ≥ 1 mm in two or more contiguous electrocardiogram (ECG) leads or an infero-lateral myocardial infarction (MI) with ST segment depression of ≥ 1 mm in ≥ 2 of leads V1-3 with a positive terminal T wave.
3. TIMI Thrombus Grade ≥ 3 in the infarct related artery. In cases where TIMI Thrombus Grade is equal to 5 (i.e. TIMI 0 flow in the infarcted artery), TIMI Thrombus Grade of at least 3 has to be re-confirmed with AWI. Patients showing TIMI Thrombus Grade of less than 3 upon AWI are no longer eligible for randomization.
4. Start of intervention within 8 h of symptom onset
5. Subject is willing and able to provide informed consent prior to the intervention

Exclusion Criteria:

1. Unconscious patients
2. Infarct related artery diameter, at visual assessment, smaller than 2.5 mm
3. Presence of severely calcified plaque(s) proximal to or at the site of the culprit lesion(s)
4. Presence of extreme vessel tortuosity proximal to or at the site of the culprit lesion(s)
5. Women of child-bearing potential (e.g. below 55 years of age, who have not undergone tubal ligation, ovariectomy or hysterectomy and last menstruation within the last 12 months)
6. Stent thrombosis as culprit lesion
7. Previous myocardial infarction in the same territory (i.e. same target vessel)
8. Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Infarct size | three days post intervention
  size assessed by measurements of creatine kinase

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Cardiocentro Ticino, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No